CLINICAL TRIAL: NCT03534908
Title: Nonalcoholic Fatty Liver Disease and Cardiovascular Disease: the Correlation Analysis and Risk Prediction Model Study
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Wuhan University (Other)
Responsible Party: Principal Investigator, Hongliang Li, MD,PhD, Wuhan University
Other Study IDs: WDRY2017-K009
Record Dates: First submitted 2018-05-11; First posted 2018-05-23 (Actual); Last update posted 2019-10-08 (Actual); Status verified 2019-10

CONDITIONS: NAFLD; Cardiovascular Diseases
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- NAFLD group: those with NAFLD
- Control group: those without NAFLD

SUMMARY:
Nonalcoholic fatty liver disease (NAFLD) is the most common cause of chronic liver disease in the world. NAFLD is associated with a lot of comorbidity, such as diabetes, metabolic syndrome, coronary heart disease and chronic kidney diseases. However, the correlation between the NAFLD and cardiovascular disease (CVD) events remains controversial. This study is an observational study based on a big retrospective cohort in china to explore the prevalence of NAFLD in China, the risk factors associated with NAFLD, as well as whether patients with NAFLD are more prone to experience CVDs and CVD events.

ELIGIBILITY:
Inclusion Criteria:

* males or females aged 18-75

Exclusion Criteria:

* malignancy except primary liver cancer
* pregnancy or breastfeeding
* liver diseases of other etiology including hepatitis C virus infection ,autoimmune hepatitis,Wilson's disease,hemachromatosis,drug-induced hepatitis,parenteral nutrition
* excessive alcohol consumption
* cases missing crucial data

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People who have taken medical examination and health checkup in the health management centers of hospitals in China.
Sampling Method: Non-Probability Sample
Enrollment: 5000000 (Estimated)
Dates: Start 2017-09-25 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
the prevalence of NAFLD in China | June，2020

SECONDARY OUTCOMES:
the risk factors associated with NAFLD | August，2020
to indicate the prevalence of CVDs and CVD events in people with and without NAFLD | October，2020

CONTACTS AND LOCATIONS:
Overall Officials: Hongliang Li, MD,PhD, Principal Investigator — Wuhan University
Locations (1):
- Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided